CLINICAL TRIAL: NCT03553758
Title: Electroencephalogram Studies of Induction and Recovery From Ketamine-Induced General Anesthesia
Brief Title: EEG Studies of Ketamine General Anesthesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018P000417
Record Dates: First submitted 2018-04-05; First posted 2018-06-12 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine (Experimental): 15 subjects undergoing ketamine general anesthesia.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Subjects' brain waves will be monitored by EEG recording under ketamine general anesthesia over the course of approximately 60 minutes. Patients pain and dissociation will be assessed before the induction of ketamine and periodically after. Approximately 1 hour after ketamine induction, Midazolam will be administered to reduce patient dissociation.

SUMMARY:
We are doing this research study to find out how and where ketamine acts in the brain. Ketamine is an anesthetic (a drug or agent used to decrease or eliminate the feeling of pain by putting you in an unconscious state). We will look at the brain using a machine that records the brain's electrical activity, called an electroencephalogram (EEG). We will assess how it impacts patient's pain responses.

DETAILED DESCRIPTION:
In this trial, participants will be given ketamine at a high enough dosage to induce general anesthesia. EEG recording will be conducted during this time. Cognitive assessments and pain monitoring will be administered at various points before and after ketamine induction.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 45
* Normal body weight and habitus, BMI less than or equal to 30
* Non-smoker
* American Society of Anesthesiologists (ASA) physical status classification P1

Exclusion Criteria:

* Cardiovascular: myocardial infarction, coronary artery disease, peripheral vascular disease, arrhythmia, congestive heart failure, valvular disease, hypertension
* Respiratory: bronchitis, chronic obstructive pulmonary disease, smoking, shortness of breath
* Hepatic: hepatitis, jaundice, ascites
* Neurologic: seizure, stroke, positive neurologic findings on neurologic examination, multiple sclerosis, Meniere's disease, Parkinson's disease, neuropathy, peripheral stenosis
* Gastrointestinal: esophageal reflux, hiatal hernia, ulcer
* Endocrine: diabetes, thyroid disease
* Renal: acute or chronic severe renal insufficiency
* Hematologic: blood dyscrasias, anemia, coagulopathies, on anticoagulant therapy
* Musculoskeletal: prior surgery or trauma to head neck or face, arthritis, personal or family history of malignant hyperthermia
* Psychiatric: history or treatment for an active psychiatric problem, depression
* Reproductive: pregnancy, breast-feeding
* Medications: regular use of prescription and non-prescription medications expected to affect CNS function, St. John's Wort
* Allergies: labetalol, ondansetron, glycopyrrolate, ketamine, midazolam

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 16
Completed Screening Visit | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 1 patient was enrolled in the study, but did not complete any study activities.
Arm/Group | Ketamine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity Pre- and Post-Ketamine Induction
Description: Average Pain Intensity prior to ketamine induction, 30 minutes post ketamine, 60 minutes post ketamine, 75 minutes post ketamine, and 120 minutes post ketamine. PROMIS Pain Intensity 1a was used to assess pain delivered by a pre-calibrated pain cuff. Scale of 0 (no pain) to 10 (worst imaginable pain).
Time Frame: Approximately 125 minutes
Population: 1 patient did not complete assessments after recovery of responsiveness.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ketamine EEG Dynamics: 15 subjects undergoing ketamine general anesthesia.
  Subjects' brain waves will be monitored by EEG recording under ketamine general anesthesia over the course of approximately 60 minutes. Patients pain and dissociation will be assessed before the induction of ketamine and periodically after. Approximately 1 hour after ketamine induction, Midazolam will be administered to reduce patient dissociation.
Arm/Group | Ketamine EEG Dynamics
Number analyzed (Participants) | 14
score on a scale
  Pre-Ketamine | 7.9 (0.5)
  30 minutes Post-Ketamine | 1.6 (1.6)
  60 minutes Post-Ketamine | 4.1 (2.2)
  75 minutes Post-Ketamine | 4.3 (2.2)
  120 minutes Post-Ketamine | 5.4 (2.3)

2. Secondary Outcome: Average Dissociation States Score Pre- and Post-Ketamine Induction
Description: Patients were assessed for dissociation states prior to the induction of ketamine and at 60 minutes, 75 minutes, and 120 minutes after Ketamine was administered. The Clinician Administered Dissociation States Scale was used to measure dissociation. Each section is scored 0 (not at all) to 4 (extreme), and totaled. The minimum total score is 0 (best, no dissociation at all) and the maximum total score is 92 (worst, the most dissociation).
Time Frame: About 125 minutes
Population: 1 patient did not perform assessments after recovery of responsiveness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 14
score on a scale
  Pre-Ketamine | 0.2 (0.4)
  60 minutes post-ketamine | 22.1 (17)
  75 minutes post-ketamine | 14.3 (11.6)
  120 minutes post-ketamine | 5.2 (7.3)

3. Secondary Outcome: Difference of the Mean Clinician Administered Dissociative States Scale Before and After Midazolam Administration
Description: Midazolam was administered approximately 60 minutes after the administration of Ketamine in order to reduce the effects of Ketamine on dissociation. Dissociation was measured using the Clinician Administered Dissociative States Scale. Each section is scored 0 (not at all) to 4 (extreme), and totaled. The minimum total score is 0 (best, no dissociation at all) and the maximum total score is 92 (worst, the most dissociation). The difference of the mean Clinician Administered Dissociative States Scale before and after Midazolam administration was found.
Time Frame: About 60 minutes
Population: 1 patient did not complete assessments after recovery of responsiveness.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 14
score on a scale | 10.3 [3.4 to 17.1]

ADVERSE EVENTS:
Time Frame: From initiation of anesthesia during the first study visit to completion of the study visit, which was approximately 2 hours.
Description: Adverse events and other events were determined by regular investigator assessment and self-reporting.
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT03553758/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03553758/Prot_SAP_001.pdf